CLINICAL TRIAL: NCT06776016
Title: A Prospective, Single-Arm, Single-Center Study of Dietary Supplements in the Treatment of Radiation-Induced Rectal Injury
Brief Title: Dietary Supplements to Treat Radiation-Induced Rectal Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP202402
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Radiotherapy; Radiation Proctitis
Keywords: radiotherapy; radiation proctitis; tributyrin; rectal bleeding; butyrate
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Butyrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary supplements (Experimental): Participants receive dietary supplements combined with supportive care.
  Interventions: Dietary Supplement: Butyrate

INTERVENTIONS:
Dietary Supplement: Butyrate — Agent: The dietary supplement contains tributyrin, a pro-drug of butyrate. Method: Participants receive the supplement orally at a dose of 20 ml, 2-3 times daily, 12 weeks.

SUMMARY:
This clinical study is a prospective, single-arm, single-center trial aimed at assessing the safety and efficacy of tributyrin (TB) as dietary supplements in the treatment of chronic radiation-induced rectal injury (RRI). We hypothesize that these supplements will help improve rectal bleeding symptoms and elevate the quality of life for patients. The study will test whether the supplements can lower the LENT-SOMA scales of rectal bleeding and enhance overall patient health. Efficacy will be evaluated through blood tests and other non-invasive methods, ensuring patient safety and comfort throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* At least 3 months since the completion of pelvic radiotherapy
* No evidence of tumor recurrence or metastasis
* Rectal bleeding with grade 1-2 by LENT-SOMA scales

Exclusion Criteria:

* Acute or chronic infectious diseases
* Serious systemic diseases
* Known allergies to any components of the study medication
* Colonoscopy indicating rectal ulceration (>1cm2), fistula, stricture, or necrosis
* Late complications related to pelvic radiation injury
* Other hemorrhagic or coagulation disorders
* Previous rectal resection
* Bowel obstruction or perforation that require surgery
* Cognitive or psychological disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with alleviated rectal bleeding (degraded by 1 or more) | At the time of 12 weeks since the start of treatment
  The symptom of rectal bleeding will be assessed by LENT-SOMA scales

SECONDARY OUTCOMES:
Number of participants with mild rectal bleeding (grade 0-1) | At the time of 24 weeks since the start of treatment
  The symptom of rectal bleeding will be assessed by LENT-SOMA scales

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China